CLINICAL TRIAL: NCT01639118
Title: Prospective Observational Cohort Study Of A Size Tailored Approach To Repair Umbilical And Epigastric Primary Ventral Hernias
Brief Title: Prospective Study Of A Size Tailored Approach To Repair Umbilical And Epigastric Primary Ventral Hernias
Acronym: SITUP
Status: Terminated | Type: Observational
Why Stopped: Perception of an increased incidence of C-Qur V-patch mesh infection, with need for removal, compared to other meshes used for umbilical hernia repair.
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Stijn De Sutter, Dr. Stijn De Sutter, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: SITUP-2012
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Ventral Hernia; Umbilical Hernia; Epigastric Hernia
Keywords: primary ventral hernia repair with mesh; umbilical hernia repair; epigastric hernia repair; C-Qur V-patch; Size tailored repair; preperitoneal repair; abdominal hernia; dual sided mesh
MeSH Terms: conditions — Hernia, Ventral; Hernia, Umbilical; Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary ventral hernias, such as umbilical and epigastric hernias, are best repaired with abdominal wall reinforcement by mesh implantation. Mesh-devices using a dual-sided mesh technology have been developed for the specific indication of small ventral hernias; this technique is very attractive because the mesh can be introduced through a nearly invisible scar in the umbilicus. The dual layer of the mesh inhibits the formation of adhesions of the viscera to the mesh so, if wanted, it can be positioned in a intraperitoneal position. No literature is available on the adequate size of mesh needed to repair a hernia defect of an umbilical or epigastric hernia. Very small hernias are now often enlarged for repair with a large mesh device. Small hernias might benefit of repair with a small mesh device so no enlargement of the defect is necessary Larger hernias might benefit from a larger mesh size to have more overlap of the mesh beyond the hernia defect.

With this prospective cohort study the investigators want to explore the efficacy of C-QUR V-Patch of different sizes for the different sizes of hernia defects.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients that are planned for surgical repair of a primary umbilical or epigastric hernia will be considered to enter the study.

Exclusion Criteria:

* patients refusing to participate at the follow up visits
* pregnancy
* age < 18 years
* life expectancy less than 12 months
* recurrent umbilical or epigastric hernia
* incisional or trocar site hernias
* emergency operations
* liver cirrhosis or ascites
* cancer patients
* concomitant surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stijn De Sutter, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares; Filip Muysoms, MD, Study Director — Algemeen Ziekenhuis Maria Middelares; Iris Kyle-Leinhase, PhD, Study Chair — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Oost Vlaanderen, Belgium